CLINICAL TRIAL: NCT04277208
Title: Opioid Free Arthroscopic Rotator Cuff Repair: A Prospective Observational Trial
Brief Title: Opioid-Free Study in Arthroscopic Rotator Cuff Repair
Status: Completed | Type: Observational
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Other Study IDs: 2018LAustin
Record Dates: First submitted 2019-08-05; First posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Arthroscopic Rotator Cuff Repair

SUMMARY:
The purpose of this study is to develop and test an opioid-free pain control protocol for patients undergoing arthroscopic rotator cuff repair.

ELIGIBILITY:
Inclusion Criteria:

* All patients over the age of 18
* clinically indicated for an Arthroscopic Rotator Cuff Repair (ARCR)

Exclusion Criteria:

* Patients with irreparable rotator cuff tears
* allergic or sensitivity to the study medication
* intolerance to pain protocol
* history of gastrointestinal issues
* renal disease
* any evidence of glenohumeral arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing ARCR will be asked to participate in this survey study
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2018-12-13 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Time to fulfill oxycodone prescription | within first 3 days of surgery
  data collected to the time from surgery until the patient chooses to fulfill a prescription for opioid medication following surgery

SECONDARY OUTCOMES:
VAS pain (Visual Analog Scale) | Post-operative day 3
  patient-reported pain as measured on a scale from 0-10. Zero means no pain and 10 being worst pain imaginable
Patient satisfaction | Post-operative day 3
  Patient will be asked on a 5 point likert scale to rate their satisfaction with their post-operative pain regime

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Institute, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No